CLINICAL TRIAL: NCT06298461
Title: Bowel Preparation for Colonoscopy Among Individuals With IBD: A Randomized Controlled Trial
Brief Title: Bowel Preparation for Colonoscopy Among Individuals With Crohn's and Ulcerative Colitis Disease.
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Canadian IBD Research Consortium (CIRC) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BowelPrep
Record Dates: First submitted 2024-02-06; First posted 2024-03-07 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Crohn Disease; Ulcerative Colitis
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OSS (Active Comparator)
  Interventions: Drug: KleanLyte
- 2L PEG (Active Comparator)
  Interventions: Drug: Bi-PegLyte

INTERVENTIONS:
Drug: KleanLyte — Laxative for colonoscopy bowel preparation
  Arms: OSS
Drug: Bi-PegLyte — Laxative for colonoscopy bowel preparation
  Arms: 2L PEG

SUMMARY:
The purpose of this study is to compare how effective and how tolerable two different bowel preparation laxatives are for colonoscopy. The aim is to compare oral sulfate solution (OSS) to another laxative called 2L polyethylene glycol (PEG) solution to see which is more effective and more tolerable by individuals with IBD (Crohn's disease or Ulcerative colitis).

ELIGIBILITY:
Inclusion Criteria:

1. Crohn's disease or ulcerative colitis patients scheduled or about to be scheduled for colonoscopy.
2. Age > 18 years
3. Out-patients

Exclusion Criteria:

1. Prior subtotal or total colorectal resection
2. Contraindications to use of 2L polyethylene glycol (2L-PEG) or Oral Sulfate Solution (OSS): Known renal insufficiency, congestive heart failure, cirrhosis, severe electrolyte imbalance.
3. Colonoscopy being repeated because of poor preparation in the preceding six months.
4. Allergies to the employed bowel preparations
5. Toxic megacolon, ileus, suspected or diagnosed bowel obstruction.
6. IBD patients thought to be too sick to undergo a full colonoscopy preparation in the opinion of the investigator/treating physician; hospitalized crohn's disease or ulcerative colitis patients.
7. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 418 (Estimated)
Dates: Start 2024-07-04 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Quality of bowel cleanliness | 1 year
  The primary outcome will be adequate quality of bowel cleanliness. Proportion with adequate cleansing will be measured by Boston Bowel Preparation Scale Score ≥2 in all segments.
Quality of bowel cleanliness | 1 year
  The primary outcome will be adequate quality of bowel cleanliness. Proportion with adequate cleansing will be measured by the Ottawa scale score as a binary adequate/inadequate score (≤7) will be recorded.

SECONDARY OUTCOMES:
Volume of laxative intake | 1 year
  Will compare completion of laxative intake.
Endoscopic Outcomes | 1 year
  Will compare dysplasia detection rate.
Endoscopic Outcomes | 1 year
  Will compare withdrawal time.
Endoscopic Outcomes | 1 year
  Will compare total procedure time.
Endoscopic Outcomes | 1 year
  Will compare cecal intubation rate
Patient experience data | 1 year
  Will determine the proportion of patients in each group reporting: use of split dose and day before bowel preparation (even though they were prescribed split-dose) , incontinence episodes during bowel preparation and during travel to the colonoscopy appointment; total duration of sleep; number of nocturnal awakenings: patient willingness to repeat colonoscopy using the same preparation; pre-colonoscopy anxiety rating; difficulty with bowel preparation rating. The study specific patient questionnaire will be administered prior to the colonoscopy to avoid any contamination by the experience of the colonoscopy.
Crohn's disease or ulcerative colitis flares after colonoscopy | One month
  A one month phone call to determine diagnosed flares within a month
Endoscopic Outcomes | 1 year
  Will also compare the proportion of patients requiring repeat colonoscopy because of an inadequate bowel preparation. Will collect data on mucosal abnormality suspected by endoscopist to be due to bowel preparation.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared.